CLINICAL TRIAL: NCT06975215
Title: Pre-emptive Coil Embolization in Endovascular Aortic Repair: The PRIZE Study
Brief Title: Pre-emptive Coil Embolization in Endovascular Aortic Repair
Acronym: PRIZE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRIZE
Record Dates: First submitted 2025-05-05; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Aneurysm; Endovascular Aortic Repair; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVAR (Active Comparator): EVAR, as per standard of care
  Interventions: Procedure: EVAR
- EVAR + embolization (Experimental): EVAR, as per standard of care, associated with concomitant embolization
  Interventions: Device: Concomitant embolization; Procedure: EVAR

INTERVENTIONS:
Device: Concomitant embolization — This will include EVAR, following the standard pathway of care, associated with embolization. The decision to perform side-branch embolization or aneurysm sac embolization will be left to each participating centre/physician.
  Arms: EVAR + embolization
Procedure: EVAR — Endovascular aortic aneurysm repair

SUMMARY:
Abdominal aortic aneurysms are often treated with a minimally invasive procedure called endovascular aortic repair (EVAR). While EVAR is widely used, it can sometimes lead to complications over time, and some patients may require further procedures. One of the main issues is endoleak, which occurs when blood continues to flow into the aneurysm sac after treatment. This often happens because small nearby blood vessels, or other sources, continue to supply blood to the aneurysm.

A potentialy strategy to reduce the risk of endoleak is pre-emptive embolization-a technique used during EVAR to block these sources of persistent blood flow. This can include embolization of side branches, the aneurysm sac, or other contributing vessels. Early findings suggest that pre-emptive embolization may lower the risk of endoleaks, but it is still uncertain whether it improves long-term outcomes.

The PRIZE study (Randomized Controlled Trial on Pre-emptive Coil Embolization in Endovascular Aortic Repair) is designed to answer this question. In this research, patients are randomly assigned to one of two groups: one group will receive EVAR with pre-emptive embolization, and the other will receive EVAR without it.

Two main outcomes will be assessed. The first is aneurysm sac regression at two years, meaning a reduction in the size of the aneurysm sac after treatment. This is important because sac shrinkage after EVAR has been linked to lower overall mortality, even though the exact reasons for this are not yet fully understood. The second main outcome is the rate of aortic-related events over five years, as ensuring the long-term durability of treatment is a key goal of this study. Secondary outcomes, including quality of life, patient satisfaction, and cost-effectiveness will also be evaluated.

Currently, there is no clear agreement on whether pre-emptive embolization should be routinely used during EVAR. In a recent international survey, 76% of aortic specialists agreed that more evidence is needed. The PRIZE study aims to provide that evidence. If pre-emptive embolization proves effective, it could become a standard addition to EVAR, helping to improve both the immediate success and long-term durability of treatment. If not, the study will help avoid unnecessary procedures, ensuring patients receive only treatments that offer real benefits.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic aneurysms with a maximum aortic diameter above the threshold for repair level.
* High-risk criteria for type 2 endoleaks

Exclusion Criteria:

* Does not fulfill instructions for use for standard EVAR
* Contraindication for EVAR
* Life expectancy less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Aneurysm sac regression at 2 years | 24 months
  Changes in the maximum aneurysm sac volume, which will be to assessed by an independent core lab.
Rate of aortic events at 5 years | 60 months
  The number of study participants with aortic events, including:
  * Aortic-related reinterventions
  * Development of type I/III, with or without reintervention
  * Development of T2EL with sac expansion >10mm with or without reintervention
  * Graft infection
  * Aneurysm rupture
  * Aortic-related death

IPD SHARING:
Plan to Share IPD: Undecided